CLINICAL TRIAL: NCT03089853
Title: Smart Telehealth Exercise Intervention to Reduce COPD Readmissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Surya P Bhatt, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160504003
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Results first posted 2020-09-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pulmonary rehabilitation; telehealth; smart; technology; Neuromuscular Electrical Stimulation (NEMS); acute exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized controlled study where subjects will be randomized in a 2:1 ratio to either receive remote tele pulmonary rehabilitation intervention and NMES or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Subjects randomized to intervention arm will have a device applied to their thigh on either side, and subject to neuromuscular electrical stimulation for 30 minutes daily for 2 weeks, followed by pulmonary rehabilitation exercises delivered at home via a smart phone for an additional 10 weeks. Rehabilitation will involve aerobics, strength training as well as breathing exercises.
  Interventions: Device: Neuromuscular electrical stimulation (NMES)
- Usual Care Arm (No Intervention): Usual care will consist of a protocolized regimen of 5 days of systemic steroids, unless the treating physician determines a different regimen, in which case the change will be documented.

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — Bipolar self-adhesive neuromuscular stimulation electrodes will be placed over the quadriceps femoris muscle group. Stimulation pulses (30 Hz trains of 300 μsec biphasic pulses) will be delivered using the neuromuscular electrical stimulator. A 5 sec on/25 sec off work/rest ratio will be used initially, progressing to 10 sec on/30 sec off. The patient will be fully supported while knee extensions are performed as the participant sits in a chair. Current from the stimulator will be manually increased and determined by patient tolerance. The goal for each patient will be to reach the highest tolerable amplitude (up to 100mA). Training will be performed on each quadriceps femoris muscle, 30 minutes/day, for 2 weeks including hospital stay till return to the COPD Clinic. This will be followed by pulmonary rehabilitation exercises delivered at home via a smart phone for an additional 10 weeks. Rehabilitation will involve aerobics, strength training as well as breathing exercises.
  Other Names: Respond II neuromuscular electrical stimulator
  Arms: Intervention Arm

SUMMARY:
This is a prospective randomized controlled study to test the hypothesis that neuromuscular electrical stimulation (NMES) and remote pulmonary rehabilitation at home offered via a smart technology, called Smart TeleHealth, results in a reduction of systemic inflammation, via reduction of skeletal muscle tissue inflammation, and thereby improves functional capacity, and thus, reduces the rate of readmissions following hospitalization for acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD). This study will enroll up to 40 participants at the University of Alabama at Birmingham (UAB), about 30 will get Smart Telehealth and NMES, and 10 will get usual care.

DETAILED DESCRIPTION:
The overall hypothesis of our proposal is that neuromuscular electrical stimulation (NMES) and remote pulmonary rehabilitation at home offered via smart technology results in a reduction of systemic inflammation, via reduction of skeletal muscle tissue inflammation, and thereby improves functional capacity, and thus, reduces the rate of readmissions following hospitalization for acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD.) We propose the following specific aims:

Aim 1: To determine if an NMES and remote tele pulmonary rehabilitation intervention reduces 30-day all cause readmissions in patients hospitalized for acute exacerbation of COPD. Skeletal muscle dysfunction is associated with the number of hospital admissions, duration of hospital stay and total number of exacerbations. We and others have shown that applying NMES results in significant improvements in quadriceps muscle strength. It is plausible that targeting skeletal muscle dysfunction will result in improved respiratory outcomes. Based on our preliminary results comparing our exercise intervention with historic data, we hypothesize that a combination of early in-hospital and home NMES and home pulmonary rehabilitation using smart technology will prevent hospital readmissions following an acute exacerbation of COPD.

Aim 2: To evaluate the effects of an NMES and remote tele pulmonary rehabilitation intervention on muscle strength, dyspnea and respiratory quality of life in COPD post hospital discharge. Skeletal muscle dysfunction contributes to the morbidity associated with acute exacerbations, results in a longer duration of hospital stay and a shorter time to readmission, and is associated with more frequent exacerbations. We hypothesize that by preventing deconditioning, improving muscle bioenergetics and positively affecting muscle strength, NMES and home pulmonary rehabilitation will improve respiratory quality of life, dyspnea and functional capacity. We will compare outcome measures for respiratory morbidity at baseline with those at 12 weeks.

Aim 3: To evaluate the effects of NMES and remote tele pulmonary rehabilitation intervention on systemic and muscle inflammation. Acute exacerbations of COPD are associated with sustained systemic inflammation and the mechanism for this may be perpetuation of inflammation by a skeletal muscle reservoir. We have previously shown that older patients such as those with COPD are more susceptible to muscle inflammation. Based on our preliminary results showing significant benefits, we hypothesize that the reduced readmission rates are a direct effect of lowering muscle inflammation. We hypothesize that inflammation arising from the lungs is perpetuated by pro-inflammatory signaling in the skeletal muscles that sustains systemic inflammation, and this can be reduced by a combination of early NMES and exercise therapy at home by reducing skeletal muscle production of pro-inflammatory cytokines. We will perform quadriceps muscle biopsy at baseline and at 4 weeks to demonstrate reduction in pro-inflammatory signaling in skeletal muscles at 4 weeks in the intervention arm and anticipate that this reduction will be associated with reduction in systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are hospitalized with an acute exacerbation of COPD and can be enrolled within 36 hours of hospitalization.
* Age 40 years or older.

Exclusion Criteria:

* Secondary diagnosis of congestive heart failure and other respiratory conditions that could confound the diagnosis such as pneumonia, bronchiectasis and lung cancer will be excluded.
* Those on invasive or mechanical ventilation will not be enrolled.
* Participants with pacemakers/defibrillators will not be enrolled due to concern for interaction with NEMS.
* Inability to consent for themselves.
* Pregnant or breastfeeding women will be excluded to minimize the risks of neuromuscular electrical stimulation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surya P Bhatt, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care Arm
Started | 4 | 3
Completed | 2 | 2
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (2.8) | 65.3 (9.6) | 62.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of All-cause Readmissions
Description: The primary outcome is the rate of all-cause readmissions within 30 days following an index hospitalization for Chronic Obstructive Pulmonary Disease (COPD) exacerbation.
Time Frame: Up to Day 30
Population: We were unable to analyse because of the small sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Secondary Outcome: Change in Forced Expiratory Volume During First Second (FEV1)
Description: This outcome will be measured using spirometry.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Dyspnea - Modified Medical Research Council (mMRC) Score
Description: mMRC scale is a five-point scale originally published in 1959 that considers certain activities, such as walking or climbing stairs, which provoke breathlessness.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Dyspnea - San Diego Shortness of Breath Questionnaire (SOBQ)
Description: SOBQ is a self-administered questionnaire to rate the level of dyspnea associated with activities of daily living. The minimum clinically important difference (MCID) if 5 units.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in COPD Related Quality of Life - COPD Assessment Test (CAT)
Description: CAT is a self-administered questionnaire where a change of 2 units is considered clinically significant.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Muscle Strength of Quadriceps
Description: Measured using a dynamometer in pounds/kilograms.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: 30-second Chair Test to Measure Skeletal Muscle Dysfunction, Leg Strength and Endurance
Description: Scores range from 4 to 14, depending on age and sex. Higher scores indicate higher levels of functioning. MCID is 2.
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Changes in Systemic Inflammation
Description: Blood levels of C-Reactive Protein (CRP), Fibrinogen, Interleukin 6 (IL-6) and Tumour Necrosis Factor alpha (TNF-alpha)
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Changes in Muscle Inflammation
Description: Pro-inflammatory signaling in quadriceps skeletal muscle
Time Frame: 12 weeks
Population: We were unable to analyse because of the small sample size.
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Three months
Description: No adverse events were observed.
Arm/Group | Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03089853/Prot_SAP_000.pdf